CLINICAL TRIAL: NCT03615339
Title: The Use of Fermented Whey Concentrate in Healthy Adults
Brief Title: Pilot Trial Investigating Fermented Whey Supplementation in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: A. Vogel (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 799
Record Dates: First submitted 2018-06-25; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-07

CONDITIONS: Healthy
Keywords: Food supplement, Fermented food, Whey

STUDY DESIGN:
Masking Description: Unlabelled bottles of treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Molkosan (Experimental): Consumption of Molkosan (fermented whey) 20ml to be diluted in 200ml water prior to use twice a day (morning & evening).
  Total duration was 6 weeks.
  Interventions: Dietary Supplement: Molkosan

INTERVENTIONS:
Dietary Supplement: Molkosan — Twice daily (AM and PM) 20ml of fermented whey concentrate consumed diluted in 200ml water

SUMMARY:
Pilot trial: 6-week single arm intervention. Healthy adults (male and female) consume Molkosan (fermented whey) twice a day (AM & PM).

DETAILED DESCRIPTION:
Molkosan® is made from fresh organic whey using a special fermentation process involving lactic acid producing bacteria (L+ lactic acid 70g/L). The company, A.Vogel (Roggwil, Switzerland) will provide the product and we will collect biological samples for analysis in a proof of concept study design that will provide preliminary data for future larger studies.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65
* BMI 18-40 kg/m-2

Exclusion Criteria:

* Diabetes
* Severe gastrointestinal disorders,
* Kidney disease,
* Thromboembolic or coagulation disease,
* Hepatic disease,
* Alcohol or any other substance abuse
* Gout
* Eating disorders
* Unregulated thyroid disease
* Dairy intolerance
* Antibiotic use within the last 3 months, including prescribed use
* Current prebiotic or prebiotic use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-03-16 (Actual); Primary Completion 2015-07-07 (Actual); Study Completion 2015-07-07 (Actual)

PRIMARY OUTCOMES:
Change in microbiota activity | Baseline, day 21 and 42
  Faecal short-chain fatty acids, measured by gas chromatography

SECONDARY OUTCOMES:
Change in glucose tolerance (Oral glucose tolerance test (OGTT) | Baseline, day 21 and 42
  Six blood samples will be collected during the course of 3 hours (0, 30, 60, 90,120 and 180 min) using a cannulation after consuming 75 g of Polycal liquid (glucose load). Plasma glucose level and insulin are analysed as total area under the curve (AUC) and incremental AUC.

OTHER OUTCOMES:
Change in microbiota composition - 16s rRNA (ribosomal ribonucleic acid) sequencing | Baseline, day 21 and 42
  16S rRNA extracted from fresh stool samples (<16hrs)
Subjective assessment of digestion and bowel movements | Baseline and day 14-18
  Volunteer self-reported symptoms measured by questionnaire
Energy intake | Baseline and day 14-18
  4-day weighed food diary analysed for energy intake and macronutrient composition
Blood pressure | Screening, baseline and day 42
  Repeated in triplicate, measured in mmHg
Pulse | Screening, baseline and day 42
  Triplicate measurement, expressed as beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra M Johnstone, Ph.D, Principal Investigator — Rowett Institute, University of Aberdeen
Locations (1):
- The Rowett Institute, Human Nutrition Unit, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith NM, Maloney NG, Shaw S, Horgan GW, Fyfe C, Martin JC, Suter A, Scott KP, Johnstone AM. Daily Fermented Whey Consumption Alters the Fecal Short-Chain Fatty Acid Profile in Healthy Adults. Front Nutr. 2020 Sep 30;7:165. doi: 10.3389/fnut.2020.00165. eCollection 2020. PMID 33102510
- See also: A. Vogel product website and description — https://www.avogel.co.uk/food/products/molkosan-digestion/